CLINICAL TRIAL: NCT04599933
Title: A Multi-Center, Double-Masked, Vehicle-Controlled, Evaluation of the Efficacy and Safety of CSF-1 in the Temporary Correction of Presbyopia (the NEAR-1 Study: Near Eye-vision Acuity Restoration)
Brief Title: An Evaluation of the Efficacy and Safety of CSF-1 in the Temporary Correction of Presbyopia (NEAR-1)
Acronym: NEAR-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orasis Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-150-0002
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2020-10

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSF-1 (Experimental): One drop bilaterally twice daily for approximately 2 weeks.
  Interventions: Drug: CSF-1
- Vehicle (Placebo Comparator): One drop bilaterally twice daily for approximately 2 weeks.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CSF-1 — One drop bilaterally twice daily for approximately 2 weeks.
  Other Names: pilocarpine HCl 0.4%
  Arms: CSF-1
Drug: Vehicle — One drop bilaterally twice daily for approximately 2 weeks.
  Arms: Vehicle

SUMMARY:
This is a 4-visit, multi-center, randomized, double-masked, vehicle-controlled study evaluating the safety and efficacy of CSF-1 in the temporary correction of presbyopia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have presbyopia.

Exclusion Criteria:

Subjects must not:

* Have any contraindications to the study medications or diagnoses that would confound the study.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Orasis Investigative Site, Sun City, Arizona
  - Orasis Investigative Site, Glendale, California
  - Orasis Investigative Site, Los Angeles, California
  - Orasis Investigative Site, Fort Myers, Florida
  - Orasis Investigative Site, Mt. Dora, Florida
  - Orasis Investigative Site, Morrow, Georgia
  - Orasis Investigative Site, Overland Park, Kansas
  - Orasis Investigative Site, Louisville, Kentucky
  - Orasis Investigative Site, Kansas City, Missouri
  - Orasis Investigative Site, St Louis, Missouri
  - Orasis Investigative Site, Henderson, Nevada
  - Orasis Investigative Site, Elizabeth City, North Carolina
  - Orasis Investigative Site, Cranberry Township, Pennsylvania
  - Orasis Investigative Site, Wilkes-Barre, Pennsylvania
  - Orasis Investigative Site, Rapid City, South Dakota
  - Orasis Investigative Site, Memphis, Tennessee
  - Orasis Investigative Site, El Paso, Texas

REFERENCES:
- [Derived] Holland E, Karpecki P, Fingeret M, Schaeffer J, Gupta P, Fram N, Smits G, Ignacio T, Lindstrom R. Efficacy and Safety of CSF-1 (0.4% Pilocarpine Hydrochloride) in Presbyopia: Pooled Results of the NEAR Phase 3 Randomized, Clinical Trials. Clin Ther. 2024 Feb;46(2):104-113. doi: 10.1016/j.clinthera.2023.12.005. Epub 2024 Jan 11. PMID 38216351

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CSF-1 | Vehicle
Started | 155 | 154
Completed | 146 | 147
Not Completed | 9 | 7
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Screen Failure | 1 | 2

BASELINE CHARACTERISTICS:
Population: The subject demographics and characteristics presented are for the Full Analysis Set (FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | CSF-1 | Vehicle | Total
Number analyzed (Participants) | 155 | 154 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (4.56) | 54.5 (4.88) | 54.7 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 92 | 185
  Male | 62 | 62 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 23 | 56
  Not Hispanic or Latino | 122 | 131 | 253
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 6 | 14 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 25 | 50
  White | 121 | 111 | 232
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 155 | 154 | 309
Iris Color [Count of Participants; unit: Participants]
  Light Iris Color | 71 | 70 | 141
  Dark Iris Color | 84 | 84 | 168
Manifest Refraction Spherical Equivalent (MRSE) [Count of Participants; unit: Participants] — Measure Description: MRSE: is the measure which allows to identify if a person is myopic (nearsighted) < -0.5D; emmetropic (normal refractive conditions) between -0.5D to <= +0.75D: or hyperopic (farsighted) >+0.75D.
  Participants
    -4.5 D to < -0.5 D | 35 | 32 | 67
    -0.5 D to <= +0.75 D | 88 | 90 | 178
    > +0.75 D to +2.0 D | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥ 3-line Gain in BDCVA (Best Distance-Corrected Visual Acuity) at 40cm and no Loss in BDCVA ≥ 5 Letters at 4m on Day 8, 1 Hour Post-Dose 1.
Description: The primary end-point was measured on Day 8, 1 hour post first CSF-1 dose, as the number of participants who are responders to the treatment.
  A responder was defined as as subject with a ≥ 3-line gain in BDCVA (Best Distance-Corrected Visual Acuity) at 40cm and no loss in BDCVA ≥ 5 letters at 4m.
Time Frame: Baseline (Day 1) to Day 8 (1 hour post-Dose 1)
Population: Full analysis set (FAS): included all randomized subjects who received at least 1 dose of the study drug. Subjects in the FAS were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1 | Vehicle
Number analyzed (Participants) | 155 | 154
Participants | 60 | 26
Statistical Analysis 1: Comparison: CSF-1 vs Vehicle; All treatment comparisons for primary and secondary endpoints related to BDCVA were conducted with a logistic regression model including fixed effects of baseline BDCVA at 40 cm as a covariate and treatment; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 2.916, 95% CI 2-sided [1.663 to 5.113]

2. Secondary Outcome: Percentage of Subjects With a ≥ 3-line Gain in BDCVA at 40cm and no Loss in BDCVA ≥ 5 Letters at 4m on Day 8 at 2 Hours Post-Dose 1
Description: The key secondary endpoints were measured on Day 8 at different time points and were the percentage of subjects with a ≥ 3-line (15-letter) gain, from baseline, in BDCVA at 40 cm (Precision Vision Chart) and no loss in BDCVA ≥ 5 letters (ETDRS chart at 4 m) in the study eye.
Time Frame: Baseline (Day 1) to Day 8 (2 hours post-Dose 1)
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1 | Vehicle
Number analyzed (Participants) | 155 | 154
Participants | 61 | 26
Statistical Analysis 1: Comparison: CSF-1 vs Vehicle; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 3.035, 95% CI 2-sided [1.736 to 5.305]

3. Secondary Outcome: Percentage of Subjects With a ≥ 3-line Gain in BDCVA at 40cm and no Loss in BDCVA ≥ 5 Letters at 4m on Day 8 at 1 Hour Post-Dose 2
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Day 8 (1 hour post-Dose 2; Dose 2 occurs 2 hours following Dose 1)
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1 | Vehicle
Number analyzed (Participants) | 155 | 154
Participants | 74 | 24
Statistical Analysis 1: Comparison: CSF-1 vs Vehicle; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 4.751, 95% CI 2-sided [2.694 to 8.379]

4. Secondary Outcome: Percentage of Subjects With a ≥ 3-line Gain in BDCVA at 40cm and no Loss in BDCVA ≥ 5 Letters at 4m on Day 8 at 2 Hours Post-dose 2
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Day 8 (2 hours post-Dose 2; Dose 2 occurs 2 hours following Dose 1)
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1 | Vehicle
Number analyzed (Participants) | 155 | 154
Participants | 60 | 23
Statistical Analysis 1: Comparison: CSF-1 vs Vehicle; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 3.422, 95% CI 2-sided [1.923 to 6.090]

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | CSF-1 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/155 | 1/154
Other Adverse Events (participants affected / at risk) | 17/155 | 3/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSF-1 (N=155) | Vehicle (N=154)
Enteritis (Gastrointestinal disorders) | 0 | 1 (1) — One (0.6%) SAE of enteritis was reported in the Vehicle group, which required hospitalization. The subject was discontinued from the study after Day 26, and the event was resolved at the time of discontinuation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CSF-1 (N=155) | Vehicle (N=154)
instillation site pain (General disorders) | 9 | 1
headache (Nervous system disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT04599933/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04599933/SAP_001.pdf